CLINICAL TRIAL: NCT05658718
Title: Effects of Different Pupil Size Under Light and Dark Conditions on Nighttime Symptoms After Refractive Surgery.
Brief Title: Factors Influencing Nocturnal Symptoms After Refractive Surgery.
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Second Affiliated Hospital of Nanchang University (Other)
Responsible Party: Principal Investigator, Yifeng Yu, Deputy chief physician of Ophthalmology center of the Second Affiliated Hospital of Nanchang University, Second Affiliated Hospital of Nanchang University
Other Study IDs: [2021] No. (113).
Record Dates: First submitted 2022-11-20; First posted 2022-12-21 (Actual); Last update posted 2023-09-07 (Actual); Status verified 2023-09

CONDITIONS: Refractive Surgery; Visual Quality
Keywords: refractive surgery; glare; pupil; visual quality; Aberrations
MeSH Terms: interventions — Refractive Surgical Procedures

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- glare group.: Patients subjectively complained about glare and Binoptometer examination showed poor visual quality in dark environments, and they were classified as the glare group.
  Interventions: Procedure: refractive surgery
- non-glare group: The patients did not complain of glare and the Binoptometer examination showed good visual quality in a dark environment, and they were classified as the non-glare group.
  Interventions: Procedure: refractive surgery

INTERVENTIONS:
Procedure: refractive surgery — refractive surgery

SUMMARY:
By comparing the parameters of the two groups of patients with glare at night after refractive surgery and those without glare at night, the influence of preoperative related parameters on postoperative glare was analyzed.

ELIGIBILITY:
Inclusion criteria：

* Age ≥18 years old；
* Stable diopter (diopter change less than 0.5D in the past 2 years);
* Best corrected distance visual acuity (CDVA) of 1.0 or better；
* Anterior chamber depth (ACD) ≥2.8 mm;
* Corneal endothelial cell density (ECD) ≥ 2 000 cells/mm.

Exclusion criteria:

* History of ocular trauma or surgery;
* Suspected keratoconus;
* Previous history of other ocular diseases such as corneal inflammation or edema, glaucoma, uveitis, retinal detachment, macular degeneration, cataract, amblyopia, etc.;
* History of severe dry eye；
* Patients with systemic diseases, such as hyperthyroidism or autoimmune diseases; or severe mental disorders, such as anxiety and depression.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: People undergoing refractive surgery.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2021-11-01 (Actual); Primary Completion 2023-12-01 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
Changes of diopter under bright and dark pupils. | Preoperative
  Use OPDScan Ⅲ to measure the parameters of both eyes
Changes of diopter under bright and dark pupils. | Day 7
  Use OPDScan Ⅲ to measure the parameters of both eyes.
Changes of diopter under bright and dark pupils. | Month 1
  Use OPDScan Ⅲ to measure the parameters of both eyes.
Changes of diopter under bright and dark pupils. | Month 3
  Use OPDScan Ⅲ to measure the parameters of both eyes.
Changes of diopter under bright and dark pupils. | Month 6
  Use OPDScan Ⅲ to measure the parameters of both eyes.
objective visual quality. | Day 7
  Measurement of objective visual quality using Binopotometer.
objective visual quality. | Month 1
  Measurement of objective visual quality using Binopotometer and NIDEK Automatic computerized optometry instrument（ARK-1s).
objective visual quality. | Month 3
  Measurement of objective visual quality using Binopotometer.
objective visual quality. | Month 6
  Measurement of objective visual quality using Binopotometer.
subjective visual quality | Day 7
  Using visual quality questionnaire to evaluate patients' subjective visual quality.
subjective visual quality | Month 1
  Using visual quality questionnaire to evaluate patients' subjective visual quality.
subjective visual quality | Month 3
  Using visual quality questionnaire to evaluate patients' subjective visual quality.
subjective visual quality | Month 6
  Using visual quality questionnaire to evaluate patients' subjective visual quality.
ICL Vault | Day 7
  Measuring ICL vault with Pentacam
ICL Vault | Month 1
  Measuring ICL vault with Pentacam
ICL Vault | Month 3
  Measuring ICL vault with Pentacam
ICL Vault | Month 6
  Measuring ICL vault with Pentacam

CONTACTS AND LOCATIONS:
Locations (1):
- The Second Affiliated Hospital of Nanchang University, Nanchang, Jiangxi, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Xiong J, Xu J, Zhou M, Liu J, Wang Q, Yin X, Deng Y, Luo X, Wang N, Gui F, Yu K, Liu J, Zhu Z, Cheng C, Yu Y. Mesopic pupil indices as potential risk factors for glare disability after intraocular implantable collamer lens implantation: prospective study. J Cataract Refract Surg. 2024 Jun 1;50(6):565-571. doi: 10.1097/j.jcrs.0000000000001420. PMID 38350161